CLINICAL TRIAL: NCT00850603
Title: Safety and Immunogenicity of Intradermal, and Low-dose Subcutaneous vs Subcutaneous Administration of Menomune® - A/C/Y/W-135
Brief Title: Safety and Immunogenicity of Intradermal Versus Subcutaneous Doses of Menomune®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MPT01
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Results first posted 2009-04-30 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Meningococcal Infections; Meningitis
Keywords: Menomune® - A/C/Y/W-135; Meningococcal Infections; Meningitis
MeSH Terms: conditions — Meningococcal Infections; Meningitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 (Active Comparator): 0.5 mL Subcutaneous arm (Menomune® )
  Interventions: Biological: Meningococcal Polysaccharide Groups A\C\Y\W-135 Combined
- Group 2 (Experimental): 0.1 mL Subcutaneous arm (Menomune®)
  Interventions: Biological: Meningococcal Polysaccharide Groups A\C\Y\W-135 Combined
- Group 3 (Experimental): 0.05 mL Intradermal arm (Menomune®)
  Interventions: Biological: Meningococcal Polysaccharide Groups A\C\Y\W-135 Combined
- Group 4 (Experimental): 0.1 mL Intradermal arm (Menomune®)
  Interventions: Biological: Meningococcal Polysaccharide Groups A\C\Y\W-135 Combined
- Group 5 (Experimental): 0.15 mL Intradermal arm (Menomune®)
  Interventions: Biological: Meningococcal Polysaccharide Groups A\C\Y\W-135 Combined

INTERVENTIONS:
Biological: Meningococcal Polysaccharide Groups A\C\Y\W-135 Combined — 0.5 mL, Subcutaneous
  Other Names: Menomune® - A/C/Y/W-135
  Arms: Group 1
Biological: Meningococcal Polysaccharide Groups A\C\Y\W-135 Combined — 0.1 mL, Subcutaneous
  Other Names: Menomune® - A/C/Y/W-135
  Arms: Group 2
Biological: Meningococcal Polysaccharide Groups A\C\Y\W-135 Combined — 0.05 mL, Intradermal
  Other Names: Menomune® - A/C/Y/W-135
  Arms: Group 3
Biological: Meningococcal Polysaccharide Groups A\C\Y\W-135 Combined — 0.1 mL, Intradermal
  Other Names: Menomune® - A/C/Y/W-135
  Arms: Group 4
Biological: Meningococcal Polysaccharide Groups A\C\Y\W-135 Combined — 0.15 mL, Intradermal
  Other Names: Menomune® - A/C/Y/W-135
  Arms: Group 5

SUMMARY:
The objective of this trial is to study the administration of the Menomune vaccine given intradermally and low-dose subcutaneously versus standard subcutaneously. This study will describe the immunogenicity of Menomune® - A/C/Y/W-135 administered subcutaneously (standard dose) versus intradermally over a dose range (1/10th, 2/10th, and 3/10th of standard dose) and a low dose (2/10th of standard dose) subcutaneously.

The secondary objective is to describe the safety of the subcutaneous (SC) and intradermal (ID) routes at different dosages

DETAILED DESCRIPTION:
This trial will provide a proof of concept that a dose range of Menomune given ID can induce an immune response that is comparable to standard dosing by the SC route, and is equivalent or superior to a low dose given SC.

Subjects will be randomized according to a computer-generated randomization schedule to receive the vaccine by SC injection or by ID injection at different dosages.

ELIGIBILITY:
Inclusion Criteria :

* 18 to 55 years of age.
* Willing to return for 3 follow-up visits and comply with a 30 day follow-up period.
* Signed an informed consent form.

Exclusion Criteria :

* Allergy to any component of the vaccine and latex.
* Known or suspected immunodeficiency or receipt of immunosuppressive therapy or blood products within the previous two months.
* History of serious chronic diseases (such as cardiac or renal disease).
* Acute febrile illness at the time of visit.
* Pregnancy.
* Receipt of any vaccine within the 28 days prior to enrollment.
* Receipt of meningococcal vaccine (example in Military) within the past 5 years or history of meningococcal disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2002-10; Primary Completion 2003-05 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc
Locations (1):
- East Stroudsburg, Pennsylvania, United States

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 15 through 16 October 2002 in 1 US site
Pre-assignment Details: A total of 170 participants that met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- 0.5 mL Subcutaneous Menomune®: Participants received 0.5 mL Subcutaneous Menomune®
- 0.1 mL Subcutaneous Menomune®: Participants received 0.1 mL Subcutaneous Menomune®
- 0.05 mL Intradermal Menomune®: Participants received 0.05 mL Intradermal Menomune®
- 0.1 mL Intradermal Menomune®: Participants received 0.1 mL Intradermal Menomune®
- 0.15 mL Intradermal Menomune®: Participants received 0.15 mL Intradermal Menomune®
Period: Overall Study
Arm/Group | 0.5 mL Subcutaneous Menomune® | 0.1 mL Subcutaneous Menomune® | 0.05 mL Intradermal Menomune® | 0.1 mL Intradermal Menomune® | 0.15 mL Intradermal Menomune®
Started | 34 | 34 | 34 | 34 | 34
Completed | 34 | 34 | 34 | 34 | 34
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5 mL Subcutaneous Menomune® | 0.1 mL Subcutaneous Menomune® | 0.05 mL Intradermal Menomune® | 0.1 mL Intradermal Menomune® | 0.15 mL Intradermal Menomune® | Total
Number analyzed (Participants) | 34 | 34 | 34 | 34 | 34 | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 2 | 5 | 1 | 11
  Between 18 and 65 years | 32 | 33 | 32 | 29 | 33 | 159
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.8 (9.68) | 24.3 (7.10) | 24.4 (7.64) | 24.5 (8.46) | 28.9 (12.85) | 25.6 (9.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 16 | 15 | 17 | 93
  Male | 12 | 11 | 18 | 19 | 17 | 77
Region of Enrollment [Number; unit: participants]
  United States | 34 | 34 | 34 | 34 | 34 | 170

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ≥ 4-Fold Rise in Antibody Titers
Description: Percentage of participants with a 4-fold rise in Serum bactericidal assay using baby rabbit complement (SBA-BR) antibody titers to each meningococcal serogroup from baseline to Day 28 post-vaccination.
Time Frame: Baseline to 28 days post vaccination
Population: 4-Fold rise analysis was in the per-protocol population with valid serology data
Measure: Number; unit: Percentage of participants
Arm/Group | 0.5 mL Subcutaneous Menomune® | 0.1 mL Subcutaneous Menomune® | 0.05 mL Intradermal Menomune® | 0.1 mL Intradermal Menomune® | 0.15 mL Intradermal Menomune®
Number analyzed (Participants) | 34 | 34 | 34 | 34 | 34
Percentage of participants
  Meningococcal serogroup A | 85 | 61 | 61 | 76 | 84
  Meningococcal serogroup C | 79 | 58 | 67 | 70 | 88
  Meningococcal serogroup Y | 64 | 68 | 61 | 58 | 66
  Meningococcal serogroup W-135 | 88 | 77 | 73 | 79 | 97

2. Secondary Outcome: Number and Intensity of Solicited Local and Systemic Reactions Post-vaccination.
Description: Participants with solicited local and systemic reactions and intensity within 7 days following vaccination with Menomune®
Time Frame: Day 0 to 7 days post-vaccination
Measure: Number; unit: Participants
Arm/Group | 0.5 mL Subcutaneous Menomune® | 0.1 mL Subcutaneous Menomune® | 0.05 mL Intradermal Menomune® | 0.1 mL Intradermal Menomune® | 0.15 mL Intradermal Menomune®
Number analyzed (Participants) | 34 | 34 | 34 | 34 | 34
Participants
  Any Local Reaction | 8 | 5 | 9 | 10 | 18
  Any Grade 3 Local Reaction | 0 | 0 | 0 | 0 | 0
  Any Redness | 2 | 2 | 8 | 9 | 18
  Grade 3 Redness ( ≥ 2 inchs) | 0 | 0 | 0 | 0 | 0
  Any Swelling | 0 | 1 | 4 | 5 | 10
  Grade 3 Swelling ( ≥ 2 inchs) | 0 | 0 | 0 | 0 | 0
  Any Tenderness | 6 | 4 | 1 | 1 | 3
  Grade 3 Tenderness (disabling) | 0 | 0 | 0 | 0 | 0
  Any Pain | 1 | 0 | 0 | 1 | 0
  Grade 3 Pain (disabling) | 0 | 0 | 0 | 0 | 0
  Any Systemic Reaction | 4 | 9 | 7 | 4 | 3
  Any Grade 3 Systemic Reaction | 0 | 2 | 0 | 0 | 0
  Any Fever | 0 | 0 | 0 | 0 | 0
  Grade 3 Fever (≥ 39.6 ºC) | 0 | 0 | 0 | 0 | 0
  Any Chills | 1 | 2 | 0 | 1 | 0
  Grade 3 Chills (disabling) | 0 | 0 | 0 | 0 | 0
  Any Headache | 2 | 6 | 3 | 2 | 1
  Grade 3 Headache (disabling) | 0 | 1 | 0 | 0 | 0
  Any Dizziness | 1 | 0 | 1 | 0 | 0
  Grade 3 Dizziness (disabling) | 0 | 0 | 0 | 0 | 0
  Any Malaise | 0 | 2 | 1 | 1 | 1
  Grade 3 Malaise (disabling) | 0 | 0 | 0 | 0 | 0
  Any Myalgia | 0 | 1 | 2 | 0 | 0
  Grade 3 Myalgia (disabling) | 0 | 0 | 0 | 0 | 0
  Any Nausea | 0 | 3 | 0 | 1 | 1
  Grade 3 Nausea (disabling) | 0 | 0 | 0 | 0 | 0
  Any Vomiting | 0 | 1 | 0 | 0 | 0
  Grade 3 Vomiting (≥3 episodes) | 0 | 0 | 0 | 0 | 0
  Any Diarrhea | 0 | 2 | 0 | 0 | 0
  Grade 3 Diarrhea (≥3 episodes) | 0 | 1 | 0 | 0 | 0
  Any Arthralgia | 1 | 4 | 2 | 2 | 1
  Grade 3 Arthralgia (disabling) | 0 | 0 | 0 | 0 | 0
  Any Injection site Rash | 1 | 0 | 1 | 0 | 1

3. Primary Outcome: Geometric Mean Titers (GMTs) for Each Meningococcal Serogroup at Baseline and 28 Days Post-vaccination.
Description: GMTs and their 95% confidence interval to the vaccine meningococcal serogroups at Day 0 and Day 28 post-vaccination.
Time Frame: Baseline (Day 0) and Day 28 post-vaccination
Population: Geometric mean titers were determined in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 0.5 mL Subcutaneous Menomune® | 0.1 mL Subcutaneous Menomune® | 0.05 mL Intradermal Menomune® | 0.1 mL Intradermal Menomune® | 0.15 mL Intradermal Menomune®
Number analyzed (Participants) | 34 | 34 | 34 | 34 | 34
Titers
  Meningococcal serogroup A (Day 0) | 462.4 [222.4 to 961.4] | 320.4 [127.7 to 803.8] | 267.0 [114.5 to 622.7] | 381.6 [195.7 to 743.8] | 261.6 [131.1 to 522.1]
  Meningococcal serogroup A (Day 28) | 5496.3 [3262.8 to 9258.7] | 3662.7 [2392.4 to 5607.7] | 1775.6 [1116.3 to 2824.5] | 3079.0 [2298.4 to 4124.7] | 4013.3 [2575.7 to 6253.4]
  Meningococcal serogroup C (Day 0) | 48.1 [20.1 to 115.0] | 85.1 [34.6 to 209.7] | 50.8 [20.7 to 124.4] | 53.0 [21.6 to 129.7] | 41.5 [18.8 to 91.4]
  Meningococcal serogroup C (Day 28) | 2989.0 [1475.1 to 6056.5] | 1751.3 [934.0 to 3283.8] | 1478.0 [647.4 to 3374.3] | 1307.8 [661.8 to 2584.4] | 2780.6 [1428.3 to 5413.2]
  Meningococcal serogroup Y (Day 0) | 301.3 [138.3 to 656.5] | 166.8 [73.0 to 381.5] | 164.7 [73.3 to 370.2] | 216.4 [103.8 to 451.2] | 189.0 [93.5 to 382.1]
  Meningococcal serogroup Y (Day 28) | 1883.0 [1185.2 to 2991.4] | 2002.7 [1163.3 to 3447.9] | 1390.3 [742.1 to 2604.8] | 1603.6 [1111.6 to 2313.3] | 1887.6 [1120.4 to 3180.3]
  Meningococcal serogroup W-135 (Day 0) | 32.7 [15.3 to 69.8] | 37.7 [19.0 to 74.7] | 47.7 [24.5 to 93.0] | 34.1 [16.0 to 72.8] | 19.4 [9.7 to 38.9]
  Meningococcal serogroup W-135 (Day 28) | 1374.1 [846.9 to 2229.4] | 856.3 [465.9 to 1573.8] | 1390.3 [805.1 to 2400.9] | 1307.8 [881.6 to 1940.2] | 2006.7 [1204.5 to 3343.0]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination for 28 days post-vaccination
Arm/Group | 0.5 mL Subcutaneous Menomune® | 0.1 mL Subcutaneous Menomune® | 0.05 mL Intradermal Menomune® | 0.1 mL Intradermal Menomune® | 0.15 mL Intradermal Menomune®
Serious Adverse Events (participants affected / at risk) | 0/34 | 1/34 | 0/34 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 8/34 | 9/34 | 9/34 | 10/34 | 18/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5 mL Subcutaneous Menomune® (N=34) | 0.1 mL Subcutaneous Menomune® (N=34) | 0.05 mL Intradermal Menomune® (N=34) | 0.1 mL Intradermal Menomune® (N=34) | 0.15 mL Intradermal Menomune® (N=34)
Abdominal pain NOS (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5 mL Subcutaneous Menomune® (N=34) | 0.1 mL Subcutaneous Menomune® (N=34) | 0.05 mL Intradermal Menomune® (N=34) | 0.1 mL Intradermal Menomune® (N=34) | 0.15 mL Intradermal Menomune® (N=34)
Injection site redness (General disorders) | 2 (2) | 2 (2) | 8 (8) | 9 (9) | 18 (18)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 4 (4) | 5 (5) | 10 (10)
Injection site tenderness (General disorders) | 6 (6) | 4 (4) | 1 (1) | 1 (1) | 3 (3)
Chills (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 6 (6) | 3 (3) | 2 (2) | 1 (1)
Malaise (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 2 (2) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.